Figure 1. Design of lifestyle intervention with physical activity and diet.

Date: 12 of April 2024.



Figure 2. Design of randomized controlled trial, with measurements and time plan.

Date: 12 of April 2024



Invitation



Screening



Baseline TO



Randomization

Follow-up T1 1 month



Follow-up T2 3 months



Follow-up T3 6 months

Usual care defined as written lifestyle advice

Control group (n=60)

Individualized advice and support to physical activity and diet Intervention group (n=60)



• Intervention introduction









- Body weight
- Waist-hip circumferences
- Resting energy expenditure
- Blood pressure

## All participants

- Body weight
- Body height, waist-hip circumferences
- Resting energy expenditure
- Blood pressure
- Blood samples of risk markers
- Aerobic fitness
- Muscle strength and endurance
- Physical activity (SGPALS)
- Diet (Meal-Q)
- Health-related quality of Life (EQ-5D-3L)
- Physical activity (accelerometry)
- Geospatial data (GPS)

# Time plan

Recruitment Baseline (T0) Intervention + follow-ups (T1-T3) Intervention + follow-ups (T2-T3) Analyses and dissemination

Analyses and dissemination Meetings with steering board etc. Development of long-term intervention study

Jan - Dec 2024

Jan - Dec 2025

Jan - Dec 2026



## All participants

- Body weight (primary outcome)
- Waist-hip circumferences
- Resting energy expenditure
- Blood pressure
- Blood samples of risk markers
- Aerobic fitness
- Muscle strength and endurance
- Physical activity (SGPALS)
- Diet (Meal-Q)
- Health-related quality of Life (EQ-5D-3L)
- Physical activity (accelerometry)
- Geospatial data (GPS)

## Intervention group

Feasibility:

- Process evaluation
- Perceived barriers and facilitators for behavioral change